CLINICAL TRIAL: NCT03454633
Title: A Comparative Study of Mild Hypothermic Circulatory Arrest Versus Moderate Hypothermic Circulatory Arrest on Aortic Surgery.
Brief Title: A Comparative Study of Different Hypothermic Circulatory Arrest Strategies on Aortic Surgery.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Xiaoping Fan. MD (Other)
Collaborators: Jie He.MD (Unknown); Shihao Cai.MD (Unknown); Wenda Gu.PhD (Unknown); Haijiang Guo.PhD (Unknown); Liang Hong. MD (Unknown); Ruixing Fan.PhD (Unknown); Jingsong Huang.PhD (Unknown); Tucheng Sun.MD (Unknown); Jihai Peng.MD (Unknown)
Responsible Party: Sponsor-Investigator, Xiaoping Fan. MD, Chief Physician, Guangdong Provincial People's Hospital
Organization: Guangdong Provincial People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017316H
Record Dates: First submitted 2018-02-25; First posted 2018-03-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Morality; Hypothermic Circulatory Arrest Time; Aortic-cross Clamping Time; Cardiopulmonary Bypass Time; Operation Time; Re-Thoracotomy; ICU Stay; Mechanical Ventilation Time; Blood Transfusion; Neurological Disorder; Dialysis; Aneurysm; Endoleak; Hospital Stay
Keywords: Hyperthermic circulatory arrest; Surgery
MeSH Terms: conditions — Nervous System Diseases; Aneurysm; Endoleak

STUDY DESIGN:
Intervention Model Description: A randomised controlled study
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mild hypothermia (Experimental): Initiation of circulatory arrest using the cardiopulmonary bypass at temperature 28.1 - 34 degrees Celsius
  Interventions: Procedure: the temperature of hypothermic circulatory arrest
- Moderate hypothermia (Active Comparator): Initiation of circulatory arrest using the cardiopulmonary bypass at temperature 20.1 - 28 degrees Celsius
  Interventions: Procedure: the temperature of hypothermic circulatory arrest

INTERVENTIONS:
Procedure: the temperature of hypothermic circulatory arrest — Different temperature (mild 30 degree or moderate 25 degree) employed during the hypothermic circulatory arrest on aortic surgery.

SUMMARY:
By comparing the clinical outcome of patients underwent different hypothermic circulatory arrest (mild hypothermic versus moderate hypothermic) during aortic arch surgery, this study aims to determine the optimal hypothermic circulatory arrest strategy for aortic surgery.

DETAILED DESCRIPTION:
Hypothermic circulatory arrest (HCA) is the cornerstone of aortic surgery. It provides a bloodless and still operative field. But the side effect of hypothermia also draws people's concern. With the development of surgical techniques and cardiopulmonary bypass (CPB) management, the temperature of HCA has been raised from deep hypothermia (14.1-20 degree) to moderate hypothermia (20.1-28 degree), and it has been a primary choice for many surgeons around the world. Some of surgeons still tried to push the limit and started using mild hypothermia (28.1-34 degree), and satisfactory outcome was obtained. However, the optimal temperature of HCA has not yet been determined.

In this randomized controlled study, 80 informed and consenting patients who are scheduled for total arch replacement with concomitant proximal aortic reconstruction will be randomized to mild (28.1-34 degree) or moderate (20.1-28 degree) hypothermia during circulatory arrest. Clinical outcomes of both groups will be analyzed to determine the optimal temperature for HCA.

ELIGIBILITY:
Inclusion Criteria:

1.Patients with confirmed diagnosis (i.e.aortic dissection, marfan syndrome, aortic arch aneurysm and so on), which require total aortic arch replacement.

Exclusion Criteria:

1. Preoperative heart attack or coma.
2. Patients with surgical contraindication, including but not limited to severe cardiac,pulmonary,renal or hepatic insufficiency.
3. Pre-existing heart condition or neurological disease.
4. Variation of aortic arch or its branch vessels.
5. Patient is currently on anticoagulation therapy or has other medical condition that compromises the coagulation.
6. Patient with active infection.
7. Allergy to anaesthetic or contrast agent.
8. Pregnant or lactating female.
9. Patient is already on other medical trial.
10. Other medical, psychological or socioeconomics condition determined by investigator that is not eligible for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-08-03 (Actual); Primary Completion 2020-02-15 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
Mortality | 3 months within surgery.
  In-hospital Mortality or other related death
Re-thoracotomy | Through the hospitalization, an average of 4 weeks.
  Postoperative bleeding or other conditions require re-thoracotomy
Neurological disorder | Through the hospitalization, an average of 4 weeks.
  Any neurological event occur after surgery, including transient and permanent.

SECONDARY OUTCOMES:
HCA time | During the operation
  the time of hypothermic circulatory arrest
Aorta-cross clamp time | During the operation
  the time of aortic-cross clamp
CPB time | During the operation
  the time of cardiopulmonary bypass
Operation time | During the operation
  the time of the entire surgery.
ICU stay | Through the ICU stay, an average of 1 weeks.
  the day of ICU treatment
Time of mechanical ventilation | Through the use of ventilation, an average of 3 days.
  the time of using respirator
Blood transfusion | Through the hospitalization, an average of 4 weeks.
  the number of blood product during the hospitalization, including red blood cell, platelet, plasma and so on.
Dialysis | Through the hospitalization, an average of 4 weeks.
  postoperative renal failure requiring dialysis
Hospital stay | Through the hospitalization, an average of 4 weeks.
  the time of hospitalization
Postoperative aneurysm | 1 year within the surgery
  Aortic aneurysm develope after the surgery
Postoperative endoleak | 1 year within the surgery
  Stent-graft endoleak occurs after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Fan, PhD, Study Director — Guangdong General Hosiptal; Jie He, MD, Principal Investigator — Guangdong General Hosiptal
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No